CLINICAL TRIAL: NCT04525040
Title: Experience of Using ProbioKid for Children That Often Get Sick as a Prevention for Acute Respiratory Diseases
Brief Title: ProbioKid as Prevention Among Kids With Frequent URTI
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lallemand Health Solutions (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ProbioKid study
Record Dates: First submitted 2020-08-20; First posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-07

CONDITIONS: Respiratory Tract Infections
Keywords: Frequent respiratory infection; pediatrics; probiotics
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention arm (Experimental): Children in this arm were given ProbioKid®; one capsule daily, for 6 weeks.
  Interventions: Dietary Supplement: ProbioKid®
- Pragmatic arm (Other): Children in this arm received standard of care as usual without a preventive intervention
  Interventions: Other: Pragmatic comparator

INTERVENTIONS:
Dietary Supplement: ProbioKid® — Probiokid formulation includes three probiotic strains and fructooligosaccharides.
  Arms: Intervention arm
Other: Pragmatic comparator — Standard of care as usual without a preventive intervention
  Arms: Pragmatic arm

SUMMARY:
This study was designed to evaluate the preventive efficacy of a 6-week prophylactic administration of Probiokid® on the incidence of respiratory infections and related complications in frequently sick children.

DETAILED DESCRIPTION:
The microbiota is very important for the development of the immune system in children. Lactic acid bacteria, such as Lactobacillus and Bifidobacterium, are usually administered as probiotics (defined as live microorganisms that, when administered in adequate amounts, confer a health benefit on the host). Some probiotics were shown to sustain the development of immune competency in newborns, as well as to modulate the adaptive immune response and response to infections. For example, previous research suggests that probiotics decrease the incidence of upper respiratory tract infection (URTI). Probiokid® is a commercially-available formulation that consist of probiotics (Lactobacillus helveticus, Bifidobacterium infantis, Bifidobacterium bifidum) and fructooligosaccharides. This formulation has been shown to decrease the rate of respiratory infection in children supplemented for 3 to 9 months. Therefore the aim of this clinical trial is to assess the efficacy of Probiokid® supplemented for 6 weeks on the prevention of URTI and related complications among children (aged 3 to 10 years-old) that frequently suffer of acute respiratory infections. In addition, the impact of a prophylactic intervention with Probiokid® on the number of physician visits and antibiotic courses prescribed is assessed.

ELIGIBILITY:
Inclusion Criteria:

* Age of children from 3 to 10 years,
* High frequency of acute respiratory tract infections, characterized by a resistance index more than 0.33 (i.e. ARIs more often than once every 3 months).
* Absence of other medications that affect the immune system in the treatment regimen (except for antibiotics, as per the care provider's judgment).

Exclusion Criteria:

• Chronic pathological conditions.

Ages: 3 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2016-09-14 (Actual); Primary Completion 2017-06-25 (Actual); Study Completion 2017-06-25 (Actual)

PRIMARY OUTCOMES:
Number and duration of URTI and related complications | 6 months prior to enrollment, and 6 months follow-up
  Difference between group in the change [ follow-up - baseline]

SECONDARY OUTCOMES:
Monthly incidence of URTI | 6 months after the intervention
  Comparison of monthly incidence of URTI between the two groups during follow-up
Monthly number of visits to a specialized physician | 6 months after the intervention
  Comparison of monthly number of visits to a specialized physician between the two groups during follow-up
Resistance index | 6 months prior to enrollment and 6 months after intervention
  Comparison of change in resistance index between the two groups
Individual complication diagnosed (number of cases) | 6 months prior to enrollment and 6 months after intervention
  Comparison of the number of complications diagnosed between the two groups
Number of antibiotics prescriptions | 6 months prior to enrollment and 6 months after intervention
  Comparison of the number of antibiotic courses prescribed between the two groups during follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Yu V. Marushko, MD, Principal Investigator — Bogomolets National Medical University (Kiev, Ukraine)

IPD SHARING:
Plan to Share IPD: No